CLINICAL TRIAL: NCT04958564
Title: Comparison of Interlock Nailing Versus Dynamic Compression Plating in Transverse Fractures of Tibia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: District Headquarters Teaching Hospital Sahiwal (Other)
Responsible Party: Principal Investigator, Humayun Israr, clinical professsor and dean of orthopaedics department, District Headquarters Teaching Hospital Sahiwal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DHQTHS
Record Dates: First submitted 2021-06-25; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Transverse Fracture of Shaft of Tibia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group interlock (Active Comparator): Intra medullary device used to treat tibial shaft fractures
  Interventions: Device: DCP
- group DCP (dynamic compression plate) (Active Comparator): dynamic compression plate used to treat tibial shaft fractures
  Interventions: Device: DCP

INTERVENTIONS:
Device: DCP — 1. Dynamic compression plating to compress the fracture
  2. Intramedullary device to share the load.
  Other Names: Interlock nailing

SUMMARY:
Study aims to compare two treatment modalities for treatment of transverse fractures of tibia. One is Intramedullary interlocking nail and the other is dynamic compression plate.

DETAILED DESCRIPTION:
This study is a comparison of two devices used to teat transverse fractures of tibia and these include intra medullary rod popularly known as intra medullary nail and the second is a weight bearing device know as dynamic compression plate which is fixed with screws to diaphyseal segment of bone.

ELIGIBILITY:
Inclusion Criteria:

- Patients with closed transverse tibial fractures

Exclusion Criteria:

- Patients unsuitable for surgical intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
weight bearing | 12 weeks
  when patient started to fully bear weight on affected leg after intervention

SECONDARY OUTCOMES:
time of union | 12 weeks
  time for union during which three cortices of the bone seem united radiologically

CONTACTS AND LOCATIONS:
Overall Officials: Humayun Israr, MBBS, Principal Investigator — District Headquarters Teaching Hospital Sahiwal
Locations (1):
- Orthopaedics Department ,DHQ Teaching Hospital Hospital Sahiwal, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
All data will probably be shared to fellow researchers after publication of study .